CLINICAL TRIAL: NCT00254059
Title: A Randomized Study to Compare Polysomnography With Overnight Home Oximetry and Auto - CPAP for Diagnosis and Nasal CPAP Titration in Patients With a High Probability of Obstructive Sleep Apnea.
Brief Title: A Randomized Study to Compare Polysomnography With Overnight Home Oximetry and Auto - CPAP for Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C03-0079
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2005-11-15 (Estimated); Status verified 2005-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSAHS, OSA, CPAP, polysomnography, overnight oximetry, Obstructive sleep apnea, apnea hypopnea index, AHI, Obstructive Sleep Apnea Hypopnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Microcephaly, Primary Autosomal Recessive, 6

INTERVENTIONS:
Procedure: Ambulatory diagnosis and titration with nasal CPAP using over night oxymetry and auto CPAP and vs conventional diagnosis and titration using polysomnography

SUMMARY:
This study will look at an alternative new pathway for diagnosis and treatment based on simple procedures in the patient's own home compared with the current conventional laboratory based pathway. The purpose is to determine whether all patients with OSA require the more elaborate laboratory procedures, or whether a subgroup can be managed more simply.

DETAILED DESCRIPTION:
The research question we are exploring is whether the conventional approach is better in terms of successful treatment, compliance with treatment, and quality of life. There will be 2 arms to the study. Subject will be randomly assigned to either one of the following two treatment options: 1) the conventional investigation and nasal CPAP treatment pathway comprising 2 overnight sleep studies, one for diagnosis and one for determining the required level of nasal CPAP treatment 2) experimental pathway that uses a simplified home study (overnight oximetry), together with a machine that automatically adjusts the nasal CPAP pressure to the required amount, and a careful follow-up during the first 2 weeks of treatment.

Procedures: The study protocol will require the subject to complete the following procedures which are part of routine clinical practice: History and Physical Examination by a physician, Home Oximetry (This simple test involves wearing an oxygen probe gently wrapped around subject's finger during a night's sleep to continuously measure the amount of oxygen in blood and detect obstructions of subject's breathing. The probe is easily applied by the subject and requires no supervision), Spirometry (simple non-invasive breathing test), Standardized Sleepiness Questionnaires, Orientation and Education regarding nasal CPAP therapy, and compliance monitoring, Overnight polysomnography (This is the procedure that requires subject to spend a night in the sleep laboratory with a variety of painless and non-invasive monitoring devices attached to the body. The purpose is to obtain detailed information about subject's sleep quality, breathing, heart function, and body movements during sleep. Subject will be continuously monitored by a trained technologist during this procedure.). The following procedures are not routine and subject may be required to complete some or all of them depending on which pathway assigned to. Follow-up visits to the Clinic on Days 7 and 14 of nasal CPAP treatment for adjustments of nasal CPAP pressure as required (this could also be done at home), Repeat Home Oximetry as required, Quality of Life Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years

* Residence in the Lower Mainland
* History and physical examination findings compatible with OSAHS
* Normal spirometry. (This is necessary to avoid decreased specificity of overnight oximetry attributable to underlying lung disease)
* Epworth Sleepiness Scale > 10

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Other known disorders that cause daytime sleepiness
* Requiring sedative/hypnotic medications
* Psychiatric disorder
* Life threatening co-morbidity e.g. chronic lung disease, coronary artery disease - unstable angina, recent myocardial infarction, heart failure, seizure disorder, and previous motor vehicle accident attributed to hypersomnolence
* Language barrier
* Inability to give informed consent
* Contraindication to nasal CPAP therapy
* Previous treatment of OSAHS with nasal CPAP, oral appliance therapy or corrective upper airway surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Study Completion 2004-12

PRIMARY OUTCOMES:
The primary outcome measurement will be apnea-hypopnea index (AHI) during a full night polysomnogram performed on the effective nasal CPAP pressure after 3 months of nasal CPAP therapy.

SECONDARY OUTCOMES:
1. The study will also compare CPAP pressure between the two groups after 3 months of therapy.
2. This study will compare Epworth Sleepiness Score, arousal index and sleep efficiency index between the two groups after 3 months of therapy.
3. This study will compare Sleep Apnea Quality of Life Index between the two groups after 3 months of therapy.
4. It will compare the change in Sleep Apnea Quality of Life Index from baseline to follow-up between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ryan, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Coastal Health Research Institute, Respiratory Division, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Mulgrew AT, Fox N, Ayas NT, Ryan CF. Diagnosis and initial management of obstructive sleep apnea without polysomnography: a randomized validation study. Ann Intern Med. 2007 Feb 6;146(3):157-66. doi: 10.7326/0003-4819-146-3-200702060-00004. PMID 17283346